CLINICAL TRIAL: NCT04976725
Title: Comparison of the Effectiveness of Craniosacral Therapy and Myofacial Relaxation Techniques in People Diagnosed With Migraine
Brief Title: Comparison of Craniosacral Therapy and Myofacial Relaxation Techniques in People Diagnosed With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Physical Therapist, pHd, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10354421-2021/03-13
Record Dates: First submitted 2021-04-09; First posted 2021-07-26 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Migraine Disorders
Keywords: migraine, osteopathic maniulative treatment, myofascial release, physiotherapy
MeSH Terms: conditions — Migraine Disorders | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: 75 individuals will be included in our study, including 3 groups: control group (N= 25), osteopathic manipulative technique (n= 25), myofascial relaxation group (n=25). Which group of individuals will be determined by randomizing them with closed envelope method.
  Osteopathic Manipulative Therapy and myofascial relaxation treatment applications will be applied 2 days a week, for periods of 30 min for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ostepathic manipulative treatment (Experimental): The effects of osteopathy treatment method on the migraine
  Interventions: Other: Osteopathic Manipulative Therapy
- Myofascial relaxation Treatment (Experimental): The effects of myofascial treatment method on the migraine
  Interventions: Other: Osteopathic Manipulative Therapy
- Control treatment (Experimental): Control group will have just medication treatment
  Interventions: Other: Osteopathic Manipulative Therapy

INTERVENTIONS:
Other: Osteopathic Manipulative Therapy — 75 individuals will be included in our study, including 3 groups: control group (N= 25), osteopathic manipulative technique (n= 25), myofascial relaxation group (n=25). Which group of individuals will be determined by randomizing them with closed envelope method.
  Osteopathic Manipulative Therapy and myofascial relaxation treatment applications will be applied 2 days a week, for periods of 30 min for 4 weeks.

SUMMARY:
Headache is a neurological condition that is very common all over the world and is observed at some time in life in more than 90% of society. Migraine headache, known for thousands of years, is one of the oldest diseases of humanity. The word 'hemicrania', meaning 'half of a head', is used due to unilateral pain. Approaches to treating migraine include medication, relaxation, biofeedback, living a regular life, adequate sleep, exercise, and stress management. Neck pain is especially common in migraine patients. Exercise, manual practices, electrop novelties are used to reduce musculoskeletal problems, thus reducing the effects of migraine. Myofascial relaxation techniques, which are included in the manipulative techniques in the literature, are relaxation methods performed on myofascial trigger points.Osteopathic manual therapy (OMT) , which has recently entered the literature, 19. osteopathy, developed by Andrew Taylor STILL at the end of the century, is a treatment system characterized by focusing on integrity and using it by hand to heal diseases.The study of cranial OMM kraniyum first anatomical and physiological mechanisms for the prevention and treatment of disease as a whole is concerned with the relationship of the body, including diagnostic and therapeutic methods.It is used in the treatment of somatic dysfunction of the head and other body parts. An important component of cranial Omm is the primary respiratory mechanism, which occurs as movement of the head bones, sacrum, dural membranes, central nervous system and cerebrospinal fluid. The primary respiratory mechanism is synchronous with the cranial rhythmic impulse, a 2-phase rhythmic cycle that represents a dynamic metabolic exchange with each stage of the body. This cycle is indicated as loops between 7 and 14 per minute.Fascial mobilization therapy increases energy use in segments implemented by mechanical changes.Accordingly, it helps to reduce the spasm of these layers extending fascially, to dissolve adhesions, and to increase the range of motion of the joint.

H0: Osteopathic Manipulative Therapy has no effect on migraine symptoms. H1: Osteopathic Manipulative Therapy has an effect on migraine symptoms. H2: myofascial relaxation techniques have no effect on migraine symptoms. H3: methods of Osteopathic Manipulative Therapy have an effect on migraine symptoms.

H4: myofascial relaxation techniques and osteopathic manipulative treatment methods have no superiority over each other.

H5: myofascial relaxation techniques and osteopathic manipulative treatment methods have superiority over each other.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 Diagnosed with chronic migraine Patients who have recently been diagnosed with chronic migraine who have not taken any medications so far for migraines.

Exclusion Criteria:

Those in the drug group had a decommissioning of drug use for 4 weeks Suspicion or presence of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 4 weeks , evaluation will be apply at the beginning and after treatment
  Pain severity: the visual Analog scale (VAS) will be used to determine the pain severity of cases during rest and activity, the cases will be divided into 10 equal parts of 100 mm and the number values placed between 0 and 10 on the horizontal line will be described. "I don't have any pain" was announced as 0 points, "unbearable pain" was announced as 10 points, "moderate pain" was announced as 5 points. They will be asked to mark one of the values in accordance with these descriptions
24-Hour Daily Life Scale In Migraines | 4 weeks , evaluation will be apply at the beginning and after treatment
  The validity and reliability of the "24-hour migraine quality of life scale", developed to determine changes in their quality of life within 24 hours after the first dose of the migraine drug they received after the onset of migraine headache, was examined for Turkish society.
Migraine Disability Index | 4 weeks , evaluation will be apply at the beginning and after treatment
  MIDAS is a scale that has been developed to measure headache-related yeti loss and to improve patient-doctor communication about the functional consequences of migraine.
Corbin Posture Analysis | 4 weeks , evaluation will be apply at the beginning and after treatment
  Anterior, posterior and lateral posture analysis of individuals Corbin posture analysis will be performed. Anterior tilt of the head, rounded back, shoulder protraction, kyphosis, lordosis, abdominal sagging, Genu recurvatum, lateral tilt of the head, protrusion of the scapula and scoliosis will be evaluated
Cranial Analysis | 4 weeks , evaluation will be apply at the beginning and after treatment
  The presence of asymmetry on the face will be evaluated together with parallel lines passing through the eyes, nose and lip on the face
Cervikal Range of Motion | 4 weeks , evaluation will be apply at the beginning and after treatment
  Cervical region normal joint movement (NEH), cervical region extension, rotation, flexion and lateral flexion motion angles will be measured with universal goniometer.
Trigger Point Palpation | 4 weeks , evaluation will be apply at the beginning and after treatment
  The trigger point in the chewing and neck muscles will be investigated by fingertip palpation in a stretched muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanyaaku, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
YES

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/J.JCM.2019.12.001
- See also: Related Info — http://www.biomedcentral.com/1472-6882/8/28
- Available data/document: Statistical Analysis Plan — https://doi.org/10.1016/J.JCM.2019.12.001